CLINICAL TRIAL: NCT00504361
Title: Collection of Blood for Gene Expression Study in Individuals With Chronic Lung Diseases (Qatar)
Brief Title: Blood Collection From Individuals With Lung Disease for Genetic Studies (Qatar)
Acronym: Q-BC
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other); Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 0605008516; HMC RC#373/2006 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Asthma; COPD; Interstitial Lung Disease; Cystic Fibrosis; Lung Cancer
Keywords: Asthma; COPD; Interstitial Lung Disease; Cystic Fibrosis; Lung Cancer; smokers; non-smokers
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Cystic Fibrosis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This protocol is designed to collect a small amount of blood for extraction of DNA (genetic material) for the study of the genetic basis of lung disease. Genomic DNA will be extracted, and genome wide SNP analysis and promoter sequences for genes will be obtained. The goal is to find single nucleotide polymorphims (SNP), small changes in single genes that affect disease risk, to see if they correlate with lung disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Lung Disease: Individuals with at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-ray consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; (6) patients with diseases of organs with known association with lung disease; and (7) individuals suspected of history of lung diseased based on history and/or physical examination
- 2: Normal Control: Individuals without a history of lung disease.

SUMMARY:
This is a research study where researchers are collecting blood to evaluate the genetic characteristics of individuals with chronic lung diseases, including asthma, COPD (chronic obstructive pulmonary disease), interstitial lung disease, cystic fibrosis, and lung cancer. The investigators hope to be able to identify an association between a genetic make-up in the blood samples and the risks of developing a particular lung disease, or severity of a lung disease. The findings of this study might be important to develop future preventative methods and potential treatments for the management of lung disease.

DETAILED DESCRIPTION:
This protocol is designed to collect a small amount of blood for extraction of DNA (genetic material) for the study of the genetic basis of lung disease. The study population will include individuals with known lung diseases and controls without lung disease. Individuals in the study population will be individuals at the Hamad Medical Corporation, Qatar (HMC), as well as other individuals recruited for this study. In this protocol, researchers will survey medical records of patients with chronic lung disease, in order to study the clinical characteristics of these individuals, and the researchers will collect blood to evaluate the genetic characteristics of individuals with chronic lung diseases including asthma, and COPD (chronic obstructive pulmonary disease), pulmonary fibrosis, and lung cancer. The researchers will also collect blood samples of individuals without lung disease to serve as control.

This protocol, to be carried out at Weill Cornell Medical College - Qatar and Hamad Medical Corporation, Qatar, parallels a similar approved protocol IRB #0508008095, entitled, "Collection of Blood for Gene Expression/Genomic Studies in Individuals with Chronic Lung Diseases", ongoing at Weill Cornell Medical College - New York.

ELIGIBILITY:
Lung Disease group. Individuals with lung disease who fit the following criteria will be enrolled.

Inclusion criteria

* Must provide informed consent
* Males and females, age 18 years and older
* Evidence of lung disease proven by at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-rays and/or chest CT consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) diseases of organs with known association with lung disease; and (7) individuals suspected of history of lung diseased based on history and/or physical examination

Exclusion criteria

* Individual refuses consent.

Normal control group. For the purpose of this protocol, "normal" will include individuals without history of chronic lung disease, including asthma, and without recurrent or recent (within 3 months) acute pulmonary disease, and will be determined by the following criteria:

Inclusion Criteria:

* Must provide informed consent.
* Males or females ages 18 years and older.
* Non-smokers, ex-smokers and smokers.

Exclusion Criteria:

* Individual refuses consent.
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals visiting the Medicine Department at the Hamad Medical Corporation, Qatar for standard clinical care will be recruited.
  Controls will be obtained from volunteers without a history of lung disease. Family members of patients may be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Genomic DNA will be extracted, and genome wide SNP analysis and promoter sequences for genes will be obtained. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Cornell Medical College, NY and Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided